CLINICAL TRIAL: NCT02737085
Title: the Sequential Therapy of CD19-targeted and CD20-targeted CAR-T Cell Therapy for Diffuse Large B Cell Lymphoma(DLBCL)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Jieping Chen, Head of Hematology Department, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Southwest Hospital, China
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-03

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: CD19-targeted CAR-T Cell; CD20-targeted CAR-T Cell; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diffuse Large B Cell Lymphoma(DLBCL) (Experimental): The trial will be conducted in a manner of simon two-stage design with Anti-CD19 CAR-T cells and Anti-CD20 CAR-T cells, beginning in the first stage with the aim of over 30% reaction rate among 15 patients with Diffuse Large B Cell Lymphoma(DLBCL). Only when the expected reaction rate is achieved the 30 patients left can be recruited.
  Interventions: Biological: Anti-CD19 CAR-T cells and Anti-CD20 CAR-T cells

INTERVENTIONS:
Biological: Anti-CD19 CAR-T cells and Anti-CD20 CAR-T cells — Patients receive autologous-derived CD19-targeted CAR-T cells following CD20-targeted CAR-T cells after receiving lymphodepleting chemotherapy.
  Other Names: CD19-targeted CAR-T cells and CD20-targeted CAR-T cells

SUMMARY:
The main purpose of this study is to explore the sequential therapeutic effect of CD19-targeted and CD20-targeted chimeric antigen receptor T(CAR-T) cells in the treatment of Diffuse Large B Cell Lymphoma(DLBCL)

DETAILED DESCRIPTION:
The anti-CD20 antibody has been broadly used in the treatment of B cell malignancies and exhibited good clinical outcomes. The CD19-targeted CAR-T has shown excellent therapeutic efficiency in B cell malignancies,especially in acute lymphocytic leukemia. However, patients treated with CD19-targeted CAR-T may face relapse of CD19 mutation. Therefore we attempt to treat Diffuse Large B Cell Lymphoma(DLBCL) patients by sequential therapy of the 2 targets and hope to combine their advantages.

ELIGIBILITY:
Inclusion Criteria:

1. CD19-expressing and CD20-expressing Diffuse Large B Cell Lymphoma(DLBCL) must be assured and must be relapsed or refractory disease after at least one standard chemotherapy and one salvage regimen. According to current traditional therapies, there must be no available alternative curative therapies and subjects must be either ineligible for allogeneic stem cell transplant (SCT), have refused SCT, or have disease activity that prohibits SCT at this time.
2. Patients enrolled must have an evaluated score above 60 with KPS.
3. Expected survival time of patients enrolled is over 3 months.
4. Gender is not limited, age from 14 years to 75 years.
5. Patients must have measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
6. Patients are expected to survive for more than 3 months by their physicians at the time of enrollment.
7. Adequate absolute CD3 count estimated need to be assured for obtaining target cell dose based on dosage cohorts.
8. Subjects with the following CNS status are eligible only in the absence of neurologic symptoms suggestive of CNS leukemia, such as cranial nerve palsy: CNS 1, defined as absence of blasts in cerebral spinal fluid (CSF) on cytospin preparation, regardless of the number of WBCs; CNS 2, defined as presence of < 5/uL WBCs in CSF and cytospin positive for blasts, or > 5/uL WBCs but negative by Steinherz/Bleyer algorithm CNS3 with marrow disease who has failed salvage systemic and intensive IT chemotherapy (and therefore not eligible for radiation)
9. Patients with isolated CNS relapse will be eligible if they have previously been treated with cranial radiation (at least 1800 cGy).
10. Ability to give informed consent.
11. Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus.
12. Cardiac function: Left ventricular ejection fraction greater than or equal to 40% by MUGA or cardiac MRI, or fractional shortening greater than or equal to 28% by ECHO or left ventricular ejection fraction greater than or equal to 50% by ECHO.
13. Renal function: Creatinine level of peripheral blood is required no greater than 133umol/L.
14. Patients with history of allogeneic stem cell transplantation are eligible if there is no evidence of active GVHD and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
15. Patients volunteer to participate in the research

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for participation in the study:

1. Patients are evaluated below 50 scores with KPS.
2. Evident signs suggesting that patients are potentially allergic to cytokines.
3. Frequent infection history and recent infection is uncontrolled.
4. Patients with concomitant genetic syndrome: patients with Down syndrome, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome
5. Active acute or chronic graft-versus-host disease (GVHD) or requirement of immunosuppressant medications for GVHD within 4 weeks of enrollment.
6. Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. For additional details regarding use of steroid and immunosuppressant medications.
7. Pregnancy and nursing females. HIV infection.
8. Active hepatitis B or active hepatitis C.
9. Participation in a prior investigational study within 4 weeks prior to enrollment or longer if required by local regulation. Participation in non-therapeutic research studies is allowed.
10. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
11. Patients with a known history or prior diagnosis of other serious immunologic, malignant or inflammatory disease.
12. Other situations we think not eligible for participation in the research.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events That Are Related to Treatment | 2 years
  Determine the toxicity profile of the CD19-targeted and CD20-targeted CAR-T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jieping Chen, MD,PhD, Principal Investigator — Department of Hematology, Southwest Hospital, Third Military Medical University
Locations (1):
- Southwest Hospital of Third Millitary Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338